CLINICAL TRIAL: NCT02575027
Title: 4π Radiotherapy for Recurrent Glioblastoma Multiforme: A Feasibility Trial
Brief Title: Palliative 4pi Radiotherapy in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-001086; NCI-2015-01449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-001086 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH)
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma; Recurrent Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (4pi radiotherapy) (Experimental): Patients undergo 4pi radiation simulation and planning followed by 5 to 10 daily fractions of 4pi palliative radiotherapy. If an acceptable plan cannot be achieved using 4pi planning, then the patient will be treated with standard radiation therapy planning for palliative re-irradiation.
  Interventions: Radiation: Palliative Radiation Therapy; Other: Questionnaire Administration; Radiation: Radiation Therapy Treatment Planning and Simulation

INTERVENTIONS:
Radiation: Palliative Radiation Therapy — Undergo 4pi palliative radiotherapy
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy Treatment Planning and Simulation — Undergo 4pi radiation simulation and planning
  Other Names: Radiation Therapy Treatment Planning/Simulation

SUMMARY:
This pilot clinical trial studies the feasibility of palliative 4pi radiotherapy in treating patients with glioblastoma multiforme that has come back after standard chemoradiation. A new radiotherapy delivery planning system, called 4pi radiotherapy, may help improve radiation delivery by improving dose coverage to the treatment target, while reducing the dose to surrounding normal tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the accuracy of dose delivery and patient comfort with treatment time.

II. To evaluate normal tissue dose volume statistics and compare to standard planning.

OUTLINE:

Patients undergo 4pi radiation simulation and planning followed by 5 to 10 daily fractions of 4pi palliative radiotherapy. If an acceptable plan cannot be achieved using 4pi planning, then the patient will be treated with standard radiation therapy planning for palliative re-irradiation.

After completion of study treatment, patients are followed up at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary glioblastoma multiforme (GBM)
* Patient must have previously undergone standard chemoradiation- 59.4 Gy (1.8 Gy/fraction) or 60 Gy (2.0 Gy/fraction) with concurrent and adjuvant Temodar (temozolomide)
* Patient must be diagnosed with recurrent GBM either with biopsy or radiographically
* Karnofsky Performance Status (KPS) >= 70
* Ability to understand and willingness to sign a written informed consent
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented; women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study treatment and for up to 4 weeks following the study treatment

  * For the purpose of this study, all women are considered to be of childbearing potential unless they are post-menopausal at least 1 year since last menses), biologically sterile, or surgically sterile (i.e. hysterectomy, bilateral oophorectomy or tubal ligation)

Exclusion Criteria:

* Patients with active infection
* Patients with KPS < 70 and/or unable to tolerate potentially longer treatment times
* Refusal to sign informed consent
* Pregnant women, or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception for the entire study period and for up to 4 weeks after the study treatment
* Note: Concurrent and/or adjuvant chemotherapy does not make a patient ineligible; participation in a concurrent treatment protocol does not make a patient ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of dose delivery | Up to 6 weeks
  The accuracy of dose delivery by 4pi will be compared to standard procedures. Standard quality assurance (QA) procedures will be employed to validate the delivery accuracy of 4pi. Specifically, a MatriXX phantom will be employed to measure the dose in both the coronal and sagittal planes and compared to calculation. Patients with QA results showing gamma passing rates (using 3% and 3 mm dose difference and distance to agreement criteria, respectively) less than 90% in either plane or a maximum single gamma value greater than 2 will not be treated until the source of error is corrected.
Normal tissue dose volume | Up to 6 weeks
  Statistics will be compared between 4pi and standard planning. Specifically, dose to organs-at-risk (OAR) and planning target volume (PTV) coverage will be compared to assess for improved OAR sparing and improved PTV coverage with 4pi planning.
Patient comfort with treatment time, determined by a patient-completed questionnaire completed at the end of each fraction | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Tania Kaprealian, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States